CLINICAL TRIAL: NCT06552117
Title: ElastoMRI Evaluation of Hepatic Metastases in Colorectal Cancer
Brief Title: ElastoMRI Evaluation of Hepatic Metastases in Colorectal Cancer ( MetaIRM)
Acronym: MetaIRM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: APHP220209
Record Dates: First submitted 2024-07-30; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer With Liver Metastases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- immediately resectable patients. (Other): 10 immediately resectable patients receiving preoperative chemotherapy based on Folfox alone.
  Interventions: Other: an elastoMRI sequence
- potentially resectable patients (Other): 30 potentially resectable patients (borderline) with two groups of patients representing the usual combinations of triplets: chemotherapy and targeted therapy: Folfox + bevacizumab (15 patients) and Folfox + Cetuximab (15 patients).
  Interventions: Other: an elastoMRI sequence
- unresectable patients (Other): 10 unresectable patients with two groups of patients representing the usual combinations: pure cytotoxics vs cytotoxics + targeted therapy ( bevacizumab or Cetuximab).
  Interventions: Other: an elastoMRI sequence

INTERVENTIONS:
Other: an elastoMRI sequence — Addition of an MRI elasto sequence performed during MRI performed as part of the treatment

SUMMARY:
Currently, the tumor response of operated colorectal liver metastases is assessed by histology of the resection specimen.The histological data make it possible to define categories (responder, partial responder, non-responder).

Overall survival (OS: overall survival) after surgery crucially depends on the response to neoadjuvant chemotherapy. Current criteria for predicting histological response in preoperative imaging are not satisfactory.

The working hypothesis is that it is possible to better differentiate the tissue response to conventional chemotherapies and anti-angiogenics through MRI elastography by quantifying the changes in tissue mechanical properties induced by systemic treatments.

The objectives is to evaluate the mechanical properties obtained by elasto MRI according to the systemic treatments envisaged: conventional chemotherapy such as Folfox or combined with targeted therapy

DETAILED DESCRIPTION:
Currently, the tumor response of operated colorectal liver metastases is assessed by histology of the resection specimen.The histological data make it possible to define categories (responder, partial responder, non-responder).

Overall survival (OS: overall survival) after surgery crucially depends on the response to neoadjuvant chemotherapy. Current criteria for predicting histological response in preoperative imaging are not satisfactory.

The working hypothesis is that it is possible to better differentiate the tissue response to conventional chemotherapies and anti-angiogenics through MRI elastography by quantifying the changes in tissue mechanical properties induced by systemic treatments.

The objectives is to evaluate the mechanical properties obtained by elasto MRI according to the systemic treatments envisaged: conventional chemotherapy such as Folfox or combined with targeted therapy

This is an open, non-randomized, non-comparative trial with three parallel groups

* 10 patients immediately resectable and receiving preoperative chemotherapy based on Folfox alone.
* 30 potentially resectable patients (borderline) with two groups of patients representing the combinations usual triplets: chemotherapy and targeted therapy: Folfox+bevacizumab (15 patients) and Folfox + Cetuximab (15 patients).
* 10 unresectable patients with two groups of patients representing the usual combinations: cytotoxic pure vs cytotoxic + targeted therapy (bevacizumab or Cetuximab).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years old, followed for colorectal cancer with hepatic metastases.

The diagnosis of metastasis can be made: either by tumor biopsy or by the appearance during follow-up of colorectal cancer of at least one liver lesion with the characteristics of metastasis (fibrous tumor type imaging)

* Patient with an indication to receive first-line chemotherapy for liver metastases, whether or not associated with targeted therapy
* Patient with at least one hepatic metastasis greater than 2cm

Exclusion Criteria:

* Patients not affiliated with social security
* Pregnant or breastfeeding women
* Patients under guardianship, curatorship or safeguard of justice
* Patients with a contraindication to MRI or to the injection of contrast agent in MRI. The classic contraindications for MRI are defined by the French Society of Radiology:http://www.sfrnet.org/sfr/professionnels/1-fiche-information-patients/irm/index.phtml
* Lack of signed patient consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate elasticity obtained by elasto MRI according to the systemic treatments selected: conventional purified type Folfox or associated with a targeted therapy | 6 months
  The Primary endpoint is variation in the measurement of the elasticity of the metastases by elastography-MRI between the baseline MRI and the follow-up MRI according to the morphological response criteria RECIST1.1
Evaluate elasticity obtained by elasto MRI according to the systemic treatments selected: conventional purified type Folfox or associated with a targeted therapy | 6 months
  The Primary endpoint is variation in the measurement of the elasticity of the metastases by elastography-MRI between the baseline MRI and the follow-up MRI according to the morphological response Chun criteria
Evaluate viscosity obtained by elasto MRI according to the systemic treatments selected: conventional purified type Folfox or associated with a targeted therapy | 6 months
  The Primary endpoint is variation in the measurement of the viscosity of the metastases by elastography-MRI between the baseline MRI and the follow-up MRI according to the morphological response criteria RECIST1.1
Evaluate viscosity obtained by elasto MRI according to the systemic treatments selected: conventional purified type Folfox or associated with a targeted therapy | 6 months
  The Primary endpoint is variation in the measurement of the viscosity of the metastases by elastography-MRI between the baseline MRI and the follow-up MRI according to the morphological response Chun criteria

SECONDARY OUTCOMES:
Correlate in operated patients the mechanical properties obtained by elastomeric MRI with the histological response. | by preoperative
  Measurement of the elasticity and viscosity of the metastases by preoperative elastography-MRI according to the histological response classified as complete response, partial response (viable tissue less than 50% of the tumor volume), or non-responder (viable tissue greater than 50% of the tumor volume).
Compare the metastases detected of liver MRI with liver CT | Preoperative for the group of resectable patients and after 4 cycles for the potentially resectable and unresectable groups
  Number of metastases detected
Compare the type of tumor response of liver MRI with liver CT | Preoperative for the group of resectable patients and after 4 cycles for the potentially resectable and unresectable groups
  type of tumor response using RECIST 1.1
Compare tumour response of liver MRI with liver CT | Preoperative for the group of resectable patients and after 4 cycles for the potentially resectable and unresectable groups
  Chun criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gael Goujon, Principal Investigator — APHP

IPD SHARING:
Plan to Share IPD: Undecided